CLINICAL TRIAL: NCT04913779
Title: Study to Evaluate the Safety and Effectiveness of an Immunobiological Drug (Anti SARS-CoV-2) in the Treatment of Coronavirus Disease 2019 (CoViD-19)
Brief Title: Safety and Effectiveness of an Immunobiological Drug in CoViD-19
Acronym: INPB001
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Administracion Nacional de Laboratorios e Institutos de Salud Dr. Carlos G. Malbran (Other Government)
Responsible Party: Principal Investigator, Guillermo Alberto Keller, Physician. Specialist in internal medicine and clinical pharmacology, Administracion Nacional de Laboratorios e Institutos de Salud Dr. Carlos G. Malbran
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INPB001; PRIISA.BA 2578 (Registry Identifier: PRIISA.BA); RENIS IS003268 (Registry Identifier: RENIS); DI-2021-2196-APN-ANMAT#MS (Other: Disposición ANMAT)
Record Dates: First submitted 2021-06-01; First posted 2021-06-04 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: COVID-19 Pneumonia; COVID-19 Respiratory Infection; Covid19
Keywords: Anti-SARS-CoV-2; Purified F(ab')2 Fragments; Passive immunotherapy; Equine Serum
MeSH Terms: conditions — COVID-19 | interventions — Immunization, Passive; Control Groups

STUDY DESIGN:
Intervention Model Description: This is an adaptive phase 2/3, randomized, blinded, placebo-controlled study. 200 total patients (ratio 1:1) will be included with intermediate evaluations when reaching the initial 20 patients (initial analysis of safety and pharmacokinetics), 100 (analysis of safety and efficacy) and 200 (final analysis).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-SARS-CoV-2 (Active Comparator): Administration of 10 ml of a concentrated equine hyperimmune serum solution with neutralizing activity of SARS-CoV-2 not less than1/5120, administered in slow intravenous infusion (10 ml diluted in100 ml of physiological solution, administered over 50 to 60 minutes in slow drip), produced by ANLIS-Malbrán, administered twice (time 0 when incorporated into the study -initial dose- and at 48 hours -second dose-).
  Interventions: Drug: Anti-SARS-CoV-2
- Placebo (Placebo Comparator): Administration of 10 ml of a control-solution with no-neutralizing activity of SARS-CoV-2, administered in slow intravenous infusion (10ml diluted in 100 ml of physiological solution, administered over 50 to60 minutes in slow drip), produced by ANLIS-Malbrán, administered twice (time 0when incorporated into the study -initial dose- and at 48 hours -second dose-).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anti-SARS-CoV-2 — Purified F(ab')2 Fragments of Equine hyperimmune Serum with anti-SARS-CoV-2 neutralizing activity (titer 1/5120 or higher)
  Other Names: Purified F(ab')2 Fragments of Equine hyperimmune Serum; F(ab')2 Fragments; Passive Immunotherapy; Equine F(ab')2 Fragments; Hyperimmune Equine Serum; Treatment Group
  Arms: Anti-SARS-CoV-2
Drug: Placebo — Administration of 10 ml of a control-solution without neutralizing activity against SARS-CoV-2, administered in slow intravenous infusion (10 ml diluted in 100 ml of saline solution, administered over 50 to 60 minutes in slow drip), produced by ANLIS-Malbrán, administered twice (time 0 when incorporated into the study -initial dose- and at 48 hours -second dose-).
  Other Names: Control Group
  Arms: Placebo

SUMMARY:
The aims of this study is to analyze the efficacy and safety of a passive immunotherapy strategy using hyperimmune equine serum known as Anti-SARS-CoV-2 elaborated by the National Institute for the Production of Biologicals (ANLIS-Malbrán) as an addition to the standard therapeutic approach for hospitalized patients with COVID-19, in patients with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection aged 18 to 80 years.

DETAILED DESCRIPTION:
This is an adaptive phase II/III study that aims to analyze the efficacy and safety of a immunobiological drug (Anti SARS-CoV-2) in the treatment of CoViD-19. This treatment is a passive immunotherapy strategy developed as a purified F(ab')2 fraction of equine hyperimmune serum (Anti-SARS-CoV-2). The equine serum was generated from antigenic stimulation with the SARS-CoV-2 receptor binding domain (RBD) purified protein.

This type of product (equine hyperimmune serum F(ab')2) has been widely used in our country in the last 100 years with satisfactory results and an acceptable safety profile in the treatment of accidents with poisonous animals such as anti-loxosceles, anti -latrodectus, anti-scorpionic, and anti-phoneutria, anti-bothropic, anti-micrurus, and anti-crotalic sera, all developed by the National Institute of Biological Production (ANLIS-Malbrán) and distributed free of charge in public hospitals in the country .

In the present study, evaluates the effect and safety of this immunobiological treatment in patients with COVID-19 that require hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects over 18 years old and under 80 years old.
2. Positive results by RT-PCR for SARS CoV-2
3. Clinical picture compatible with respiratory compromise in the form of pneumonia attributed to COVID-19 (Stage 3, 4 or 5 according to the WHO scale), lasting up to 72 hours from the onset of symptoms to their evaluation to be incorporated into the study.
4. Patient with good disposition towards the study and that signs the informed consent.

Exclusion Criteria:

1. Patients with clinical disease corresponding to mild / asymptomatic forms (Absence of radiological infiltrate and risk factors, with normal auscultation and arterial saturation of oxygen (SatO2) greater than 95%)
2. Patients with clinical disease corresponding to severe forms (Severe pneumonia: presence of severity criteria (ATS / IDSA), one of two major or three minor criteria.)
3. Patients who have received other therapeutic strategies in the framework of an experimental study that make it difficult to evaluate the results obtained, including (but not limited to): convalescent plasma, lopinavir / ritonavir, hydroxychloroquine, and azithromycin.
4. Pregnant or lactating women.
5. Women of childbearing potential not using an effective contraceptive method (withdrawal, intrauterine device, or oral contraceptives).
6. History of severe anaphylactic reaction with the administration of equine plasma.
7. Patients with comorbidities that justify a risk of high mortality from causes independent of SARS-CoV-2 infection (eg, stage IV cancer)
8. Patient who does not consent to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in time needed to clinical improvement | Reached each day between day 1 and 28 post-inclusion in the study
  In subjects admitted to the general ward for active infection by SARS-CoV-2 and a clinical picture of pneumonia who receive supportive treatment recommended by the guidelines of the Ministry of Health of the Argentine Nation (Population), if slow intravenous administration of Anti SARS-CoV-2 in two doses 48 hours apart (Intervention) added to supportive treatment, compared to supportive treatment alone (patients will receive slow intravenous administration of a placebo solution in two doses 48 hours apart to maintain the "blind" as Comparator), changes the time needed to clinical improvement (Outcome), during 28 days after the assignment (Time).

SECONDARY OUTCOMES:
Change in the number of patients in each World Health Organization (WHO) Ordinal Scale Category (0 to 8 being 0 better and 8 worse) | days 7, 14 and 21 post-inclusion
  (a) Change in the number of patients in each World Health Organization Ordinal Scale Category (0 to 8 being 0 better and 8 worse), expecting a lower proportion of patients in categories 4, 5, 6, and 7 (OUTCOME - Efficacy);
Change in Mortality rate | 28 days post-inclusion
  (b) Change of all-cause mortality at day 28 (OUTCOME - Efficacy);
Change in Mechanical Ventilation Requirement rate | 28 days post-inclusion
  (c) Determination of the frequency of invasive mechanical ventilation in the total analysis period (OUTCOME - Efficacy);
Change in duration of oxygen treatment requirement | 28 days post-inclusion
  (d) Change of the duration of oxygen therapy quantified in days of oxygen therapy (OUTCOME - Efficacy);
Change in Length of Hospitalization | 28 days post-inclusion
  (e) Change of hospital length of hospitalization, quantified in days from study inclusion until hospital discharge (OUTCOME - Efficacy);
Change in frequency of nosocomial infection | 28 days post-inclusion
  (F) Change in the frequency of patients with nosocomial infection (OUTCOME - Efficacy);
Change in Lymphocyte cell count | 28 days post-inclusion
  (g) Change of absolute lymphocyte count (OUTCOME - Efficacy);
Change in viral RNA Negativization rate on nasopharyngeal swab test | 7, 14, 21, and 28 days post-inclusion
  (h) change in the proportion of patients with detected viral RNA and the viral RNA load, measured by quantitative reverse transcriptase polymerase chain reaction (RT-PCR), on day 7, 14, 21, and 28 (OUTCOME - Efficacy);
Description of adverse events type and frequency | 28 days post-inclusion
  (i) description of reported adverse events, discriminated by their severity, and classified according to MedDRA (OUTCOME - Safety).
Requirement of additional treatments for Adverse Drug reactions | 28 days post-inclusion
  (j) The number of subjects who required additional treatment as a consequence of reported adverse events in each therapeutic branch (OUTCOME - Safety)
Describe the AUC of purified F(ab')2 Anti-SARS-CoV-2 | Time 0 (Basal, prior to drug administration), hours 1, 3, 6, 24, 48, 49 and 96, days 7, 14, 21 and 28 days
  (k1) Describe area under the curve (AUC) of the active drug, based on concentrations determined in plasma samples obtained from the first 20 patients
Describe the Cmax of purified F(ab')2 Anti-SARS-CoV-2 | Time 0 (Basal, prior to drug administration), hours 1, 3, 6, 24, 48, 49 and 96, days 7, 14, 21 and 28 days
  (k2) Describe maximum plasma concentration (Cmax) of the active drug, based on concentrations determined in plasma samples obtained from the first 20 patients (at time Minute 0 min, hours 1, 3, 6, 24, 48, 49 and 96, day 7, 14, 21 and 28 days).
Describe the t1/2 of purified F(ab')2 Anti-SARS-CoV-2 | Time 0 (Basal, prior to drug administration), hours 1, 3, 6, 24, 48, 49 and 96, days 7, 14, 21 and 28 days
  (k3) Describe plasma half life (t1/2) of the active drug, based on concentrations determined in plasma samples obtained from the first 20 patients (at time Minute 0 min, hours 1, 3, 6, 24, 48, 49 and 96, day 7, 14, 21 and 28 days).
Describe the Ke of purified F(ab')2 Anti-SARS-CoV-2 | Time 0 (Basal, prior to drug administration), hours 1, 3, 6, 24, 48, 49 and 96, days 7, 14, 21 and 28 days
  (k4) Describe elimination constant (Ke) of the active drug, based on concentrations determined in plasma samples obtained from the first 20 patients (at time Minute 0 min, hours 1, 3, 6, 24, 48, 49 and 96, day 7, 14, 21 and 28 days).

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo A Keller, PhD, Principal Investigator — INPB - ANLIS Malbrán
Locations (1):
- Hospital General de Agudos Donación Francisco J. Santojanni, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Publication of the results of all data obtained is planned.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After completion of the study.
Access Criteria: By request to the Principal Investigator